CLINICAL TRIAL: NCT03730558
Title: Non-comparative Prospective Observational Cohort Study Describing the Safety and Efficacy of Aflibercept Administered in Combination With FOLFIRI After Failure Under Oxaliplatin + Anti-EGFR Therapy in the Treatment of Patients With Metastatic Colorectal Cancer in Practice Common
Brief Title: ZETA : Prospective Observational Study
Acronym: ZETA
Status: Completed | Type: Observational
Sponsor: Recherche clinique (Other)
Responsible Party: Sponsor-Investigator, Recherche clinique, Dr Laurent Mineur, Institut Sainte Catherine
Organization: Institut Sainte Catherine (Other)
Other Study IDs: ZETA 2017-A01724-49
Record Dates: First submitted 2018-01-10; First posted 2018-11-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Colon Cancer
Keywords: metastatic; colon cancer
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Combination Product: aflibercept + FOLFIRI — aflibercept + FOLFIRI

SUMMARY:
Primary objective

- Evaluate the efficacy in terms of progression-free survival (PFS) of aflibercept in combination with FOLFIRI in patients treated routinely for metastatic colorectal cancer (mCRC) after failure of treatment with oxaliplatin + EGFR.

Secondary objective

* Evaluate the efficacy of aflibercept in combination with FOLFIRI on the 2-year overall survival rate and the objective response rate.
* Evaluate the tolerance profile of aflibercept in combination with FOLFIRI.

  * Observational study, national, multicenter, cohort, prospective without intervention on the therapeutic strategy.•

DETAILED DESCRIPTION:
Inclusion criteria

* All patients expected to be treated with aflibercept in combination with FOLFIRI for a mCRC, after failure of treatment with oxaliplatin + anti-EGFR on the decision of the doctor (situation included in the framework of the MA of aflibercept) .
* Age ≥18 years
* Signature of the agreement for the collection of medical and personal data. (Patients who have received FOLFIRINOX in the first line metastatic are allowed) Note: Failure is defined as progression during or within 6 months after discontinuation of oxaliplatin

Exclusion criteria :

* Concurrent participation in a clinical trial
* Patients who have previously received anti-VEGF agents and / or aflibercept in one trial.
* Patients who received FOLFIRI in the first metastatic line.

ELIGIBILITY:
Inclusion criteria

* All patients expected to be treated with aflibercept in combination with FOLFIRI for a mCRC, after failure of treatment with oxaliplatin + anti-EGFR on the decision of the doctor (situation included in the framework of the MA of aflibercept) .
* Age ≥18 years
* Signature of the agreement for the collection of medical and personal data. (Patients who have received FOLFIRINOX in the first line metastatic are allowed) Note: Failure is defined as progression during or within 6 months after discontinuation of oxaliplatin

Exclusion criteria :

* Concurrent participation in a clinical trial
* Patients who have previously received anti-VEGF agents and / or aflibercept in one trial.
* Patients who received FOLFIRI in the first metastatic line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients expected to be treated with aflibercept in combination with FOLFIRI for a mCRC, after failure of treatment with oxaliplatin + anti-EGFR on the decision of the doctor (situation included in the framework of the MA of aflibercept) .
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of aflibercept in terms of progression-free survival (PFS) in association with FOLFIRI in patients treated in common practice for metastatic colorectal cancer (CCRM) after failure of oxaliplatin + anti-EGFR-based treatment | 2 years
  progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Sainte-Catherine, Avignon, Vaucluse
  - Institut Sainte Catherine, Avignon

IPD SHARING:
Plan to Share IPD: No